CLINICAL TRIAL: NCT04426526
Title: Efficacy of HIFEM Treatments for Strengthening and Toning of Arms, Lower Limbs and Oblique Muscles
Brief Title: HIFEM for Arms, Lower Limbs, and Oblique Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-799_600
Record Dates: First submitted 2020-05-22; First posted 2020-06-11 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Muscle Tone Increased
Keywords: muscle strengthening; muscle tone
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Biceps circumference reduction (Experimental): This arm will evaluate the clinical efficacy and safety of the high power magnet system for toning and strengthening of biceps brachii.
  Interventions: Device: BTL 799-2
- Triceps circumference reduction (Experimental): This arm will evaluate the clinical efficacy and safety of the high power magnet system for toning and strengthening of triceps brachii.
  Interventions: Device: BTL 799-2
- Lower limb circumference reduction (Experimental): This arm will evaluate the clinical efficacy and safety of the high power magnet system for toning and strengthening of muscles in lower limbs.
  Interventions: Device: BTL 799-2
- Oblique muscles toning (Experimental): This arm will evaluate the clinical efficacy and safety of the high power magnet system for toning and strengthening of oblique muscles.
  Interventions: Device: BTL 799-2

INTERVENTIONS:
Device: BTL 799-2 — High power magnet system

SUMMARY:
Evaluation of HIFEM treatments for strengthening and toning of arms, lower limbs and oblique muscles.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of the high power magnet system for toning and strengthening of arm, lower limb and oblique muscles. The study is a prospective multi-center open-label four-arm study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Implanted defibrillators, implanted neurostimulators
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Application in the head area
* Application in the heart area
* Malignant tumor
* Injured or otherwise impaired muscles
* Fever
* Pregnancy
* Sensitivity or allergy to latex
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia
* Patients after Cesarean section delivery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Changes in adipose and muscle tissue measured via ultrasound imaging | 7 months
  To determine the effectiveness of the device for strengthening and toning of arms, lower limbs and oblique muscles through changes in surrounding tissues, measured via ultrasound imaging. Using the obtained images, change in adipose and muscular tissues before and after the therapy sessions will be compared for every participant according to the study phase.

SECONDARY OUTCOMES:
Patient's satisfaction measured via questionnaires | 7 months
  To determine the patient's satisfaction with study treatment for non-invasive strengthening and toning of arms, lower limbs and oblique muscles.The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome where the level of agreement between "strongly agree" and "strongly disagree" should indicate the participant's satisfaction with the therapy.
Incidence Of Treatment-Related Adverse Events | 7 months
  To determine side effects and adverse events (AE) associated with the BTL 799-2 treatment of the arms, lower limbs and oblique muscles. Safety outcomes will include an evaluation of the treatment area to assess and evaluate the following:
  * Muscle pain
  * Temporary muscle spasm
  * Temporary joint or tendon pain
  * Local erythema or skin redness

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Plastic Surgical Associates, Fort Collins, Colorado
  - Juva Skin & Laser Center, New York, New York